CLINICAL TRIAL: NCT05755971
Title: Combination Taping in Knee Osteoarthritis
Brief Title: Therapeutic Effects of Combination Tape in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Osama Ragaa Abdelraouf Ibrahim, Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RES-2022-0230
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: combination taping; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Blinded randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Intervention providers and participants are not aware of the purpose of the study or group selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Receive combination taping in addition to conventional physiotherapy
  Interventions: Other: Combination taping
- control group (Other): Receive conventional physiotherapy
  Interventions: Other: Combination taping

INTERVENTIONS:
Other: Combination taping — Elastic and rigid tapes applied together for six weeks
  Other Names: conventional physiotherapy

SUMMARY:
Taping is a non-invasive technique that has been used for various musculoskeletal conditions, including knee OA. However, there is limited research on the effects of combination taping techniques on disability, functional capacity, and knee isokinetic torque in patients with knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common chronic condition, characterized by progressive loss of joint cartilage, leading to joint pain, stiffness, and functional disability. Knee OA is one of the most prevalent forms of OA, affecting millions of people worldwide. Various non-surgical treatment options have been reported, one of them is taping techniques. Combination taping is a unique treatment option, where two different types of taping is applied. However, there is limited research on the effects of combination taping techniques on disability, functional capacity, and knee isokinetic torque in patients with knee OA. So this study will be conducted to explore therapeutic effects in individuals who are suffering from knee OA

ELIGIBILITY:
Inclusion Criteria:

* second degree knee osteoarthritis

Exclusion Criteria:

* Sever obesity, sever osteoarthritis, history of knee surgery, allergy to the tape

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Nine weeks
  Knee disability questionnaire

SECONDARY OUTCOMES:
6 minute walk test | Nine weeks
  Functional test
Time up and go test | Nine weeks
  Functional test
Knee isokinetic torque | Nine weeks
  Muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Osama R Ibrahim, PhD, Principal Investigator — BMC; Olfat M Ali, PhD, Study Chair — BMC
Locations (1):
- Batterjee Medical College, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Available upon request